CLINICAL TRIAL: NCT00874393
Title: Early Blood Pressure Management in Extremely Preterm Infants Feasibility Pilot Study
Brief Title: Early Blood Pressure Management in Extremely Premature Infants
Acronym: ELGAN BP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICHD-NRN-0041; U10HD021364 (NIH); U10HD027880 (NIH); U10HD034216 (NIH); U10HD036790 (NIH); U10HD040492 (NIH); U10HD053089 (NIH); U10HD053124 (NIH); UL1RR025744 (NIH); UL1RR025764 (NIH); UL1RR025777 (NIH); U10HD027904 (NIH); U10HD027853 (NIH); U10HD040689 (NIH); U10HD027851 (NIH); UL1RR025008 (NIH); U10HD021373 (NIH); U10HD027856 (NIH); U10HD053109 (NIH); UL1RR024979 (NIH); U10HD053119 (NIH); UL1RR025747 (NIH); U10HD021385 (NIH); U10HD027871 (NIH); UL1RR024139 (NIH)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Hypotension; Blood Pressure
Keywords: NICHD Neonatal Research Network; Very Low Birth Weight (VLBW); Extremely Low Birth Weight (ELBW); Prematurity; Blood Pressure Management; Dopamine; Hydrocortisone
MeSH Terms: conditions — Premature Birth; Hypotension | interventions — Dopamine; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dopamine and hydrocortisone (Active Comparator): Dopamine AND hydrocortisone
  Interventions: Drug: Dopamine; Drug: Hydrocortisone
- Dopamine and placebo (Active Comparator): Dopamine AND normal saline placebo
  Interventions: Drug: Dopamine; Drug: Syringe Placebo
- Placebo and hydrocortisone (Active Comparator): Dextrose (D5W) placebo AND hydrocortisone
  Interventions: Drug: Hydrocortisone; Drug: Infusion Placebo
- Placebo and Placebo (Placebo Comparator): Dextrose (D5W) placebo AND normal saline placebo
  Interventions: Drug: Infusion Placebo; Drug: Syringe Placebo

INTERVENTIONS:
Drug: Dopamine — Dopamine
  Arms: Dopamine and hydrocortisone; Dopamine and placebo
Drug: Hydrocortisone — Hydrocortisone
  Arms: Dopamine and hydrocortisone; Placebo and hydrocortisone
Drug: Infusion Placebo — Dextrose (D5W)
  Arms: Placebo and Placebo; Placebo and hydrocortisone
Drug: Syringe Placebo — Normal saline
  Arms: Dopamine and placebo; Placebo and Placebo

SUMMARY:
This trial tests the feasibility of enrolling 60 extremely preterm infants in a randomized, double-blinded study of blood pressure management within 12 months. Eligible infants will receive an infusion drug (dopamine or a dextrose placebo) and a syringe drug (hydrocortisone or a normal saline placebo).

Enrolled infants will be randomized to receive one of the following drug pairs:

* dopamine and hydrocortisone
* dopamine and normal saline
* dextrose and hydrocortisone
* dextrose and normal saline.

In addition to the intervention above, the NRN is conducting a 6-month time-limited prospective observational study of all infants born at an NRN center between 23 and 26 weeks gestational age. All clinical decisions made for these babies will be at the discretion of the attending neonatologist/infant care team according to standard practice at each institution. Data on blood pressure management in the first 24 postnatal hours collected for each infant.

DETAILED DESCRIPTION:
Since most extremely preterm infants are critically ill in the immediate postnatal period, establishing "normal" blood pressure (BP) values is difficult. This lack of data makes deciding when to institute therapy for hypotension (low BP) challenging, leading to considerable variability in BP management in neonatal intensive care units (NICUs). Despite a lack of data on safety or efficacy, as many as 64% of extremely preterm infants receive inotropes (e.g., dopamine), and up to 12.4% of very low birthweight infants receive hydrocortisone for perceived hypotension. Since both untreated low BP and therapy provided for low BP may be harmful, the decision of whether to treat is an important issue. To date, no prospective randomized, controlled trial of BP management in this population has been performed.

This trial tests the feasibility of enrolling up to 60 extremely preterm infants in a randomized, double-blinded study of blood pressure management within 12 months. It will enroll 60 infants between 23 0/7 and 26 6/7 weeks gestational age born at 6 participating NICHD Neonatal Research Network sites. Eligible infants will receive a study infusion drug (dopamine or a dextrose placebo) and a study syringe drug (hydrocortisone or a normal saline placebo). Infants will be randomized to receive one of the following drug pairs: (1) dopamine and hydrocortisone; (2) dopamine and a placebo (normal saline solution); (3) a placebo (dextrose) and hydrocortisone; or (4) placebo (dextrose) and placebo (normal saline). (NOTE: dopamine is normally mixed with dextrose and hydrocortisone is mixed with saline solution before being administered, which is why two different placebos are being used in this trial.)

The information gathered will provide a framework for the design of a potential larger, multi-centered, randomized control trial.

NOTE: The NICHD Neonatal Research Network has received a FDA exemption from the IND regulations for this trial.

In addition to the interventional trial above, the NRN is conducting a 6-month time-limited prospective observational study of all infants born at an NRN center between 23 and 26 weeks gestational age. All clinical decisions made for these babies will be at the discretion of the attending neonatologist/infant care team according to standard practice at each institution. Data on blood pressure management in the first 24 postnatal hours collected for each infant.

Based on slow rate of recruitment, a time-limited observational study of hypotension in ELBW infants has been added to the current study.

ELIGIBILITY:
Inclusion Criteria:

* Inborn infants
* 23 0/7 to 26 6/7 weeks estimated gestational age
* Umbilical arterial catheter in place at study entry
* <= 24 hours of age

Exclusion Criteria:

* Terminally ill infants
* Infants that have received (prior to enrollment): >20 ml/kg in fluid boluses, indomethacin, or ibuprofen
* Infants with major congenital anomalies

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Enrollment and completion of 60 infants | 1 year

SECONDARY OUTCOMES:
Death | 1 week and prior to hospital discharge
Duration of antihypotensive therapy | First 96 postnatal hours
Receipt and timing of medical and/or surgical therapy for a PDA | To hospital discharge
Use of open-label antihypotensive therapies (inotropes, corticosteroids, blood and plasma volume expanders) for persistently low BP with biochemical evidence of poor perfusion | First 96 postnatal hours
Spontaneous gastrointestinal perforation | First 7 days
In-hospital complications (grade III or IV intraventricular hemorrhage, cystic periventricular leukomalacia, necrotizing enterocolitis requiring surgical intervention, retinopathy of prematurity requiring laser surgery, or bronchopulmonary dysplasia) | To hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Beau J. Batton, MD, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Ronald N. Goldberg, MD, Principal Investigator — Duke University; Krisa P. Van Meurs, MD, Principal Investigator — Stanford University; Waldemar A Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Kristi L. Watterberg, MD, Principal Investigator — University of New Mexico; Roger G. Faix, MD, Principal Investigator — University of Utah; Abhik Das, PhD, Principal Investigator — RTI International; Edward F. Bell, MD, Principal Investigator — University of Iowa; Abbot R. Laptook, MD, Principal Investigator — Brown University; Barbara J. Stoll, MD, Principal Investigator — Emory University; Brenda P. Poindexter, MD MS, Principal Investigator — Indiana University; Kurt Schibler, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Kathleen A. Kennedy, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Pablo J. Sanchez, MD, Principal Investigator — University of Texas; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; Ivan D. Franz III, MD, Principal Investigator — Tufts University
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Result] Batton BJ, Li L, Newman NS, Das A, Watterberg KL, Yoder BA, Faix RG, Laughon MM, Van Meurs KP, Carlo WA, Higgins RD, Walsh MC; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Feasibility study of early blood pressure management in extremely preterm infants. J Pediatr. 2012 Jul;161(1):65-9.e1. doi: 10.1016/j.jpeds.2012.01.014. Epub 2012 Feb 14. PMID 22336574
- [Derived] Batton B, Li L, Newman NS, Das A, Watterberg KL, Yoder BA, Faix RG, Laughon MM, Stoll BJ, Higgins RD, Walsh MC; Eunice Kennedy Shriver National Institute of Child Health & Human Development Neonatal Research Network. Early blood pressure, antihypotensive therapy and outcomes at 18-22 months' corrected age in extremely preterm infants. Arch Dis Child Fetal Neonatal Ed. 2016 May;101(3):F201-6. doi: 10.1136/archdischild-2015-308899. Epub 2015 Nov 13. PMID 26567120
- [Derived] Batton B, Li L, Newman NS, Das A, Watterberg KL, Yoder BA, Faix RG, Laughon MM, Stoll BJ, Van Meurs KP, Carlo WA, Poindexter BB, Bell EF, Sanchez PJ, Ehrenkranz RA, Goldberg RN, Laptook AR, Kennedy KA, Frantz ID 3rd, Shankaran S, Schibler K, Higgins RD, Walsh MC; Eunice Kennedy Shriver National Institute of Child Health & Human Development Neonatal Research Network. Use of antihypotensive therapies in extremely preterm infants. Pediatrics. 2013 Jun;131(6):e1865-73. doi: 10.1542/peds.2012-2779. Epub 2013 May 6. PMID 23650301
- See also: NICHD Neonatal Research Network — https://neonatal.rti.org/